CLINICAL TRIAL: NCT03309852
Title: Emergency Department Assessment of Right Ventricular Function and Size in the Post Cardiac Arrest Patient
Status: Terminated | Type: Observational
Why Stopped: Low enrollment numbers.
Sponsor: University of Manitoba (Other)
Collaborators: University of British Columbia (Other); Queen's University, Kingston, Ontario (Other)
Responsible Party: Principal Investigator, Tomislav Jelic, Assistant Professor of Emergency Medicine, University of Manitoba
Other Study IDs: B2017:104
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Right Ventricular Dysfunction; Cardiac Arrest
MeSH Terms: conditions — Ventricular Dysfunction, Right; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The right side of the heart of often overlooked in patients who are acutely unwell, as the main area of focus when performing echocardiography tends to be the left ventricle. The right ventricle can yield important diagnostic clues that can aid the clinician, particularly in cases where one may suspect elevated right sided pressures, such as those due to a pulmonary embolus. Although it is taught that a dilated right ventricle is associated in patients with pulmonary embolus, but in patients with spontaneous circulation. What is unknown is patients who sustain a cardiac arrest, does the same hold true. There is a paucity of literature surrounding the appearance of the right ventricle in the cardiac arrest patient acutely. This study aims to assess right ventricular size and function in the immediate post cardiac arrest phase.

DETAILED DESCRIPTION:
The use of point of care ultrasound (PoCUS) has grown rapidly. The incorporation of PoCUS in the assessment of patients in shock and to identify a reversible etiology to a patients cardiac arrest is widely practiced and endorsed by several organizations. While often overlooked, the right ventricle (RV) plays a critical role and often can provide clues to the etiology of a patient who is in shock. The right ventricle is very unique, as its anatomic structure, and function are markedly different then the left ventricle. What is often assessed is the size of the right ventricle. If dilated, which is defined as being >0.6 times that of the left ventricle, this could be indicative of elevated right sided pressures. In the right clinical context this may be caused by an acute pulmonary embolus. While this particular finding may raise clinical suspicion of acute right ventricular strain, point of care ultrasound cannot safely rule out acute pulmonary embolism. Several publications demonstrate the use of thrombolytics if a dilated RV is seen on PoCUS. This applies in patients with cardiac function who have not sustained a cardiac arrest. But in those patients who do sustain a cardiac arrest, these patients fall into a black hole of PoCUS findings related to the right ventricle. The international liaison committee on resuscitation has urged caution due to the unknown PoCUS findings during cardiac arrest. If one were to presume a dilated RV in a setting of a patient who sustained cardiac arrest was due to a pulmonary embolus, thrombolytics would be indicated. However, exposing the patient to thrombolytics, which in themselves carry a hemorrhage risk of 20%, is not a benign decision. Thus PoCUS findings as they pertain to the RV, in patient who sustain a cardiac arrest are unknown how they clinically correlate. Literature from critical care demonstrates that the right ventricle dilates, exhibits RV dysfunction, and carries a worse prognosis then that of the left ventricle. Recent animal data suggests that RV dilatation does occur in a porcine induced cardiac arrest model. To date, no human assessment of RV function and size in the immediate post-arrest state exists, and clearly a need to study this is evident.

objectives and hypothesis Objectives To assess the right ventricular function and size in patients who are immediately post-arrest patients.

Hypothesis Our hypothesis is that right ventricular dysfunction and dilatation is prevalent in the patients who are in cardiac arrest and in the post-cardiac arrest patient population, irrespective of they etiology of their cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Any post cardiac arrest patient who achieves return of spontaneous circulation that can have their RV assessed with point of care echo cardiography within 1 hour of ROSC.

Exclusion Criteria:

* Significant hemodynamic instability, pregnancy, incarcerated patients, age <18.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Post cardiac arrest patients.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Right ventricular dysfunction | 12 months
  Assessment of RV dysfunction in post cardiac arrest patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tomislav Jelic, MD, Principal Investigator — University of Manitoba, Health Sciences Centre
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided